CLINICAL TRIAL: NCT02859480
Title: Effectiveness and Safety of Low-dose vs. High-dose Rosuvastatin on Long-term Cardiovascular Events in Korean Patients After Percutaneous Coronary Intervention: 30-month, Prospective, Single-center, Randomized Trial
Brief Title: Dose-dependent Effect of Rosuvastatin on Long-term Clinical Outcomes After PCI
Acronym: ROSUVA-30
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hyung Joon Joo, Professor, assistant, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ED15175
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease; Coronary Disease; Cardiovascular Diseases
Keywords: Rosuvastatin Calcium; Percutaneous Coronary Intervention; Drug-Eluting Stents; Patient Outcome Assessment; Biomarkers; Hyperlipidemias; Dyslipidemias; Atherosclerosis; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Anticholesteremic Agents; Hypolipidemic Agents; Lipid Regulating Agents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Cardiovascular Diseases; Hyperlipidemias; Dyslipidemias; Atherosclerosis | interventions — Rosuvastatin Calcium; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin 5mg (Experimental): Patients are treated with Rosuvastatin 5mg/day for 30 months after percutaneous coronary intervention
  Interventions: Drug: Rosuvastatin 5mg
- Rosuvastatin 20mg (Active Comparator): Patients are treated with Rosuvastatin 20mg/day for 30 months after percutaneous coronary intervention
  Interventions: Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Rosuvastatin 5mg — Rosuvastatin 5mg tablet, q.d., for 30 months
  Other Names: Low dose group
  Arms: Rosuvastatin 5mg
Drug: Rosuvastatin 20mg — Rosuvastatin 5mg tablet, q.d., for 30 months
  Other Names: Hihg dose group
  Arms: Rosuvastatin 20mg

SUMMARY:
This study is a prospective, randomized, open-label, single-center trial designed to compare the 30 month-safety and efficacy between low-dose (5mg/dL) and high-dose (20mg/dL) rosuvastatin treatment for patients with coronary artery disease after percutaneous coronary intervention with the newer drug-eluting stent.

DETAILED DESCRIPTION:
With the development of the newer generation drug-eluting stents, percutaneous coronary intervention (PCI) has been a feasible treatment for patient with coronary artery disease. However, stent failures including in-stent restenosis and stent thrombosis have been still problematic. Moreover, neoatherosclerosis, which is the atherosclerotic process developed in the neointima within the implanted stent, has been reported to be associated with neoatherosclerotic plaque rupture and contribute to the development of acute coronary syndrome in patients after drug-eluting stent (DES) implantation.

In this perspective, recent AHA/ACC and ESC guidelines recommend the high-dose(intensity) statin therapy for patients performed PCI. However, the efficacy of the high-dose(intensity) statin therapy on cardiovascular outcomes is still controversial. Several meta-analysis failed to show the benefit of the high-dose(intensity) statin therapy to reduce the mortality. Moreover, clear evidence for the benefits of such high-dose(intensity) statin therapy has no yet been demonstrated in East Asian patients.

This trial was designed to compare the 30 month-safety and efficacy between low-dose (5mg/dL) and high-dose (20mg/dL) rosuvastatin treatment for patients with coronary artery disease after PCI in the era of the newer generation DES era.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent percutaneous coronary intervention with drug-eluting stent;

Exclusion Criteria:

* Taking other drugs which can influence the lipid profile (eg. Niacin, Fibrates;
* Serum creatinine level > 2.0 mg/dL
* Serum aspartate transaminase > 3 times upper limit of normal
* Serum alanine transaminase > 3 times upper limit of normal
* Having anaphylactic reaction for Rosuvastatin;
* Having the other contraindications for Rosuvastatin;
* Having plan to be pregnant;
* Having life expectancy less than 1 year

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular outcome | Baseline to Final visit (30 months)
  The cumulative incidences of the composite events of cardiac death, myocardial infarction, and repeat revascularization

SECONDARY OUTCOMES:
All-cause death | Baseline to Final visit (30 months)
  The cumulative incidences of all-cause death for 30 months after percutaneous coronary intervention with drug-eluting stent
Cardiac death | Baseline to Final visit (30 months)
  The cumulative incidences of cardiac death for 30 months after percutaneous coronary intervention with drug-eluting stent
Non-fatal myocardial infarction | Baseline to Final visit (30 months)
  The cumulative incidences of non-fatal myocardial infarction for 30 months after percutaneous coronary intervention with drug-eluting stent
Repeat revascularization | Baseline to Final visit (30 months)
  The cumulative incidences of any repeat coronary revascularization for 30 months after percutaneous coronary intervention with drug-eluting stent
Stent thrombosis | Baseline to Final visit (30 months)
  The cumulative incidences of stent thrombosis categorized by ARC criteria for 30 months after percutaneous coronary intervention with drug-eluting stent
Target LDL-C level achievement | 6 months of treatment and thereafter
  The percentage of the participants who reached the LDL-C level of <70mg/dL after the treatment for 6 months.
LDL-C level change | Baseline to 6 months of treatment and thereafter
  The percent changes of LDL-C level from baseline to to 6 months of treatment and thereafter
HDL-C level change | Baseline to 6 months of treatment and thereafter
  The percent changes of HDL-C level from baseline to to 6 months of treatment and thereafter
Level change of other biomarkers | Baseline to 6 months of treatment and thereafter
  The percent changes of serum level of other biomarkers from baseline to to 6 months of treatment and thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Joon Joo, MD, PhD, Principal Investigator — Department of Cardiology, Korea University Anam Hospital; Do-sun Lim, MD, PhD, Study Chair — Department of Cardiology, Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided